CLINICAL TRIAL: NCT05012761
Title: A Phase I Bridging Study to Evaluate the PK, Safety and Tolerability of SR419 in Healthy Subjects
Brief Title: The Pharmacokinetics (PK), Safety, Tolerability of SR419 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SR419-104
Record Dates: First submitted 2021-08-17; First posted 2021-08-19 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SR419 capsules (Experimental): Ascending single and multiple doses of SR419 orally
  Interventions: Drug: SR419 capsules
- Placebo (Placebo Comparator): Ascending single and multiple doses of SR419 placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SR419 capsules — Ascending single and multiple doses of SR419 orally
  Arms: SR419 capsules
Drug: Placebo — Ascending single and multiple doses of placebo orally
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I PK bridging study to evaluate the PK, safety and tolerability of SR419 in healthy subjects.

DETAILED DESCRIPTION:
The study is a Phase I study to evaluate the PK, safety, and tolerability of SR419 in healthy volunteers. The study will include 3 single-ascending-dose (SAD) cohorts and 2 multiple-dose cohorts (Part A and part B respectively), a total of 5 cohorts, and each cohort includes 3 stages: screening and baseline, treatment and safety monitoring, and safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females who are 18 to 45 years of age.
2. Based on medical history, physical examination, laboratory examination, chest X-ray, abdominal B-ultrasound, vital signs and ECG, the investigator considered that the results were normal or abnormal but no clinical significance.
3. Bodyweight of male > 50 kg, Bodyweight of female > 45 kg and body mass index (BMI) between 18 and28 kg/m2
4. Male subjects must agree to use contraception methods.
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Clinically significant history of central nervous system (CNS) disease, such as cognitive disorder and seizures. History of non-clinically significant mild anxiety (related to social stressors) or situational sleep disturbance > 6 months ago could be enrolled under the discretion of the Investigators.
2. Known history of renal dysfunction or creatinine clearance < 90 mL/min (calculated using the Cockcroft-Gault formula) at Screening.
3. Current or chronic history of liver disease or known hepatic or biliary abnormalities.
4. History of regular alcohol consumption within 6 months of screening defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~285 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits.
5. History of significant drug abuse within one year of screening or use of soft drugs (such as marijuana) within 3 months prior to screening or hard drugs (such as cocaine, methamphetamine, crack) within 1 year prior to screening.
6. History of sensitivity to any of the investigational medicinal products (IMPs), or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation.
7. History of asthma (excluding resolved childhood asthma), severe allergic responses.
8. History of hypercoagulable state or history of thrombosis.
9. A positive Hepatitis B surface antigen, positive Hepatitis C antibody and positive test for human immunodeficiency virus (HIV) antibody.
10. within 6 months of screening, Smoking more than 4 cigarettes per day (including e-cigarettes).
11. A positive drug/alcohol result at Screening or Day -1.
12. Donation or lost in excess of 500 mL of blood within 56 days of Day 1 or donation of plasma within 14 days of Day 1.
13. The subject has participated in a clinical trial within 3 months of receiving IMP.
14. Use of medication other than topical products without significant systemic absorption.
15. Unable to refrain from consumption of Seville oranges, grapefruit or grapefruit juice within 24h prior to the first dose of IMP until the Safety Follow-up visit.
16. Unable to refrain from consumption of alcohol, products containing caffeine or xanthine (such as coffee, tea, cola, chocolate) within 7 days prior to the first dose of IMP until the Safety Follow-up visit.
17. Breast-feeding and/or lactating subject.
18. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to Day 7
  Peak plasma concentration
Tmax | Up to Day 7
  Time of peak plasma concentration
AUC | Up to Day 7
  Area under the plasma concentration-time curve
CL/F | Up to Day 7
  Apparent oral clearance
t1/2 | Up to Day 7
  Terminal half-life
Rac | Up to Day 7
  Accumulation ratio

SECONDARY OUTCOMES:
The frequency and severity of AEs in healthy volunteers administrated with single and repeated oral doses of SR419 capsules | Up to Day12(+7 days) for the safety follow up since Day1
  AE: Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, Principal Investigator — Shanghai Clinical Research Center Phase I Clinical Research Unit (SCRC-PCRU)
Locations (1):
- Shanghai Clinical Research Center Phase I Clinical Research Unit (SCRC-PCRU), Shanghai, China

IPD SHARING:
Plan to Share IPD: No